CLINICAL TRIAL: NCT04717700
Title: Selinexor With Alternating Bortezomib or Lenalidomide Plus Dexamethasone in Transplant Ineligible Newly Diagnosed Multiple Myeloma Patients (SABLe): An Investigator Sponsored Trial
Brief Title: Selinexor With Alternating Bortezomib or Lenalidomide Plus Dexamethasone in TIE Newly Diagnosed MM Patients
Acronym: SABLe
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ida Bruun Kristensen (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry); Odense Patient Data Explorative Network (Other)
Responsible Party: Sponsor-Investigator, Ida Bruun Kristensen, MD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMSG 29/21
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: selinexor
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; Tablets; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- B -selinexor-lenalidomide/bortezomib-dexamethasone (Experimental): Alternating cycles of:
  Selinexor oral 40mg once weekly Lenalidomide oral 25mg d 1-21 Dexamethasone 20mg d 1+2, 8+9 and 15+16 i 28 days cycles and Selinexor oral 80mg once weekly Bortezomib sc 1.3mg/sqm once weekly Dexamethasone 20mg d 1+2, 8+9 and 15+16 in 28 days cycles for up to 16 cycles (8 of each, alternating) followed by continuos selinexor 40mg(once weekly)-lenalidomide-dexamethasone
  for up to 16 cycles followed by continuos lenalidomide-dexamethasone
  Interventions: Drug: Selinexor 20 MG Oral Tablet; Drug: Bortezomib Injection; Drug: Lenalidomide capsule; Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Selinexor 20 MG Oral Tablet — Comparing an alternating regimen of selinexor-lenalidomide/bortezomib-dexamethasone to standard bortezomib-lenalidomide-dexamethasone
  Other Names: Xpovio
Drug: Bortezomib Injection — Comparing an alternating regimen of selinexor-lenalidomide/bortezomib-dexamethasone to standard bortezomib-lenalidomide-dexamethasone
  Other Names: Velcade
Drug: Lenalidomide capsule — Comparing an alternating regimen of selinexor-lenalidomide/bortezomib-dexamethasone to standard bortezomib-lenalidomide-dexamethasone
  Other Names: Revlimid
Drug: Dexamethasone Oral — Comparing an alternating regimen of selinexor-lenalidomide/bortezomib-dexamethasone to standard bortezomib-lenalidomide-dexamethasone
  Other Names: Neofordex

SUMMARY:
An unrandomized phase 2 study of selinexor in combination with lenalidomide/ bortezomib and dexamethasone to newly diagnosed, transplant in-eligible symptomatic multiple myeloma patients in a multicenter international set-up within the Nordic Multiple Myeloma Study Group

DETAILED DESCRIPTION:
An unrandomized phase 2 study evaluating selinexor in combination with lenalidomide/ bortezomib and dexamethasone to newly diagnosed transplant in-eligible symptomatic multiple myeloma patients in a multicenter international set-up with in the Nordic Multiple Myeloma Study Group.

The study will include 50 patients, recruited within the NMSG collaborating countries. After induction patient will be treated with continued lenalidomide-dexamethasone according to SWOG, with continuous 40mg selinexor weekly in the selinexor arm (experimental arm B).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible to enroll in this study:

1. Age > 18 years
2. Willing and able to provide written informed consent in accordance with national, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of ≤ 2. ECOG 3 allowed if caused by myeloma
4. Newly diagnosed multiple myeloma with treatment demanding disease as defined by IMWG (Rajkumar, Dimopoulos et al. 2014) and measurable disease as defined IMWG 2016 criteria (Table 5) (Kumar, Paiva et al. 2016)
5. By treating physician considered in-eligible for high-dose therapy with stem-cell transplant
6. Patients must have received no prior chemotherapy for multiple myeloma. Patients must have received no prior radiotherapy to a large area of the pelvis (more than half of the pelvis). Patients must have received no prior steroid treatment for myeloma with the exception of a maximum of 14 days of treatment for symptom control (including dexamethasone 40mg).
7. Adequate hepatic function within 7 days prior to C1D1:

   1. Total bilirubin < 1.5 × upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 × ULN), and
   2. Alanine aminotransferase (ALT) normal to <2 × ULN.
8. Adequate renal function within 7 days prior to C1D1 as determined by estimated GFR of ≥ 30 mL/min, calculated using standard formula.

   1. Adequate hematopoietic function within 7 days prior to C1D1: Absolute neutrophil count ≥1000/mm3, and platelet count ≥100,000/mm3 (patients for whom <50% of bone marrow nucleated cells are plasma cells). If cytopenias are due a plasma cell infiltration in the bone marrow (biopsy-proven heavy-marrow involvement, as defined by having at least 30% marrow cellularity, with > 50% of the cells being malignant plasma cells (documented marrow results required)); in this case, although there are no required lower limits of normal for the blood counts, the treating physician must use his/her medical judgment as to the appropriateness of this study therapy for these patients.
   2. Erythropoietin-analogues are allowed.
   3. Patients must have:

      * At least a 1-week interval from the last platelet transfusion prior to the screening platelet assessment.

   However, patients may receive RBC and/or platelet transfusions as clinically indicated per institutional guidelines during the study.
9. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.
10. Patients must be able to take prophylactic anticoagulation as recommended by study
11. Patients with pathologic fractures, infection at diagnosis or symptomatic hyperviscosity must have these conditions attended to prior to registration (i.e., intramedullary rod, I.V. antibiotics, plasmapheresis)

Exclusion Criteria:

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not eligible to enroll in this study:

1. Has received selinexor or another XPO1 inhibitor previously.
2. Has any concurrent medical condition or disease (eg, uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.) that is likely to interfere with study procedures.
3. Known intolerance, hypersensitivity, or contraindication to glucocorticoids, bortezomib, lenalidomide and selinexor.
4. Pregnant or breastfeeding females.
5. Life expectancy of less than 6 months.
6. Active, unstable cardiovascular function, as indicated by the presence of:

   1. Symptomatic ischemia, or
   2. Uncontrolled clinically significant conduction abnormalities (eg, patients with ventricular tachycardia on anti-arrhythmics are excluded; patients with first degree atrioventricular block or asymptomatic left anterior fascicular block/right bundle branch block will not be excluded), or
   3. Congestive heart failure of New York Heart Association Class ≥3 or known left ventricular ejection fraction <40%, or
   4. Myocardial infarction within 6 months prior to C1D1.
7. Any active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could interfere with absorption of study treatment.
8. Inability or unwillingness to take supportive medications such as anti-nausea and anti-anorexia agents as recommended by the National Comprehensive Cancer Network® (NCCN) Clinical Practice Guidelines in Oncology (CPGO) (NCCN CPGO) for antiemesis and anorexia/cachexia (palliative care).
9. Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
10. Contraindication to any of the required concomitant drugs or supportive treatments.
11. Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Increased ORR in arm B (defined as ≥PR) at end of induction, defined according to IMWG response criteria | Estimated at 4-8 weeks after end of induction
  ORR at end of induction, with response defined according to IMWG response criteria

SECONDARY OUTCOMES:
Increased VGPR rate at end of induction in arm B | Estimated at 4-8 weeks after end of induction
  VGPR rate at end of induction
Increased rate of MRD negativity at end of induction in arm B | Estimated at 4-8 weeks after end of induction
  MRD negativity by NGS at end of induction
Decreased time to response in arm B | Estimated monthly during the first 64 weeks
  Time to at least PR from start of treatment
Evaluate toxicity rates between arm A and B, including rates of secondary primary malignancies | Estimated at 4-8 weeks after end of induction
  Comparison of toxicity rates according to NCI-CTCAE v4.03
Decreased time to at least VGPR | Estimated monthly during the first 64 weeks
  Time to at least VGPR from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ida B Kristensen, MB, Principal Investigator — Odense University Hospital; Hanne Norseth, MD, Principal Investigator — Oslo University Hospital
Locations (11):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Regionshospitalet Gødstrup, Gødstrup
  - Odense University Hospital, Odense
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- Norway (6):
  - Haukeland University Hospital, Bergen
  - Førde Central Hospital, Førde
  - Kristiansund Hospital, Kristiansund
  - Oslo Universitets Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - St. Olavs University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No